CLINICAL TRIAL: NCT00286377
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Dose Ranging Study to Evaluate the Efficacy and Safety of Prosaptide Over 6 Weeks of Treatment for the Relief of Neuropathic Pain Associated With HIV-1
Brief Title: Safety and Efficacy Study of Prosaptide to Treat Neuropathic Pain in HIV-Positive Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Savient Pharmaceuticals (Industry)
Collaborators: Neurologic AIDS Research Consortium (NARC) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C0603; NARC # 009
Record Dates: First submitted 2005-06-30; First posted 2006-02-03 (Estimated); Last update posted 2006-02-03 (Estimated); Status verified 2006-01

CONDITIONS: HIV; Peripheral Nervous System Disorders
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — prosaptide

INTERVENTIONS:
Drug: prosaptide

SUMMARY:
This is a double-blind, placebo-controlled, parallel groups study to determine whether prosptide is effective in relieving pain in patients who have sensory neuropathic pain related to their HIV infection or the drugs used to treat it.

DETAILED DESCRIPTION:
Sensory neruopathies are the most frequent neurological complicaton of HIV infection and its treatmet with antiretrovirals. To date, there are few effective treatments, and all are symptomatic treatments for pain. Management typically involves the intiation and adjustment of pain-modifying therapies, and the adjustment or discontinuation of potentially neurotoxic antiretrovirals, thereby limiting the choice of HAART regimens.

In precinical animal models,prosaptide has been shown to be efficacious in the treatment of neuropathic pain caused by a variety of different mechanisms.

Hypothesis: Prosaptide will improve neuropathic pain in HIV-associated sensory neuroathies,and will be safe and well tolerated in subjects.

Comparisons: 4, 8, or 16 mg prosaptide vs. placebo

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years and older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2003-09; Study Completion 2004-12

PRIMARY OUTCOMES:
Differnece between the pain rating at Baseline vs. Week 6 (or last week)of treatment, based on the 13-point Gracely pain intensity scale as rated by subjects and captured in an electronic diary

SECONDARY OUTCOMES:
Difference between the Beline pain rating and each week of treatment.
Number of subjects whoe were treatment successes at each week of the active treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Rehrig, MS, Study Director — Savient Pharmaceuticals, Inc.

REFERENCES:
- [Derived] Evans SR, Simpson DM, Kitch DW, King A, Clifford DB, Cohen BA, McArthur JC; Neurologic AIDS Research Consortium; AIDS Clinical Trials Group. A randomized trial evaluating Prosaptide for HIV-associated sensory neuropathies: use of an electronic diary to record neuropathic pain. PLoS One. 2007 Jul 25;2(6):e551. doi: 10.1371/journal.pone.0000551. PMID 17653259